CLINICAL TRIAL: NCT00173589
Title: Inflammatory and Fibrotic Markers and Atrial Fibrillation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700802
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-08

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
Inflammatory and Fibrotic protein markers in patients with atrial fibrillation

ELIGIBILITY:
Inclusion Criteria:

* Patients with atrial fibrillation

Exclusion Criteria:

* Patients with atrial fibrillation who are reluctant for the study

Ages: 20 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Jiunn-Lee Lin, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan